CLINICAL TRIAL: NCT01318993
Title: An Open-Label Extension Study to Assess the Safety of GSK1605786A in Subjects With Crohn's Disease
Brief Title: Open-Label Extension Study of GSK1605786A
Acronym: SHIELD-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to the lack of efficacy of GSK1605786A in Crohn's disease based on the results of Study CCX114151.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114644; 2010-022384-35 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-03-21 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease
Keywords: GSK1605786A; Inflammatory Bowel Disease; Crohn's disease; long-term treatment; quality of life; CCR9 antagonist
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — CCX282-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK1605786A (Experimental): 500 milligrams twice daily
  Interventions: Drug: GSK1605786A

INTERVENTIONS:
Drug: GSK1605786A — 500 milligrams twice daily

SUMMARY:
An open-label study to evaluate the safety and effectiveness of GSK1605786A 500 mg twice daily over 108 weeks in adult subjects with Crohn's disease. Subjects completing previous GSK-sponsored studies with GSK1605786A or subjects who withdraw early from Study CCX114157 (maintenance study of GSK1605786A) due to worsening of Crohn's disease requiring a treatment change may be eligible to participate. The primary objective is to evaluate the safety of GSK1605786A, as assessed by recording of adverse events, clinical laboratory parameters, vital signs and electrocardiogram. Secondary objectives will include assessments of effectiveness of long-term treatment with GSK1605786A. Health outcomes assessments will include changes in Inflammatory Bowel Disease Questionnaire (IBDQ), SF-36v2, EQ-5D, Work and Productivity Activity Impairment-Crohn's Disease (WPAI-CD) and receipt of disability.

DETAILED DESCRIPTION:
This is a multi-centre, open-label extension study to assess the long-term safety, tolerability and effectiveness of GSK1605786A in subjects with Crohn's disease. Subjects will enter the study via one of three routes:

1. completion of the placebo-controlled induction study, CCX114151, without achieving clinical response (CDAI decrease of at least 100 points) or clinical remission (CDAI score less than 150) at Week 12 or completion of any other GSK-sponsored induction study as designated by the sponsor
2. completion of maintenance study CCX114157 at Week 52
3. withdrawal from maintenance study CCX114157 due to worsening of Crohn's disease and requiring a treatment change.

The primary objective is to evaluate the safety of GSK1605786A, as assessed by recording of adverse events, clinical laboratory parameters, vital signs and electrocardiogram. Secondary objectives will include assessments of effectiveness of long-term treatment with GSK1605786A. Health outcomes assessments will include changes in Inflammatory Bowel Disease Questionnaire (IBDQ), SF-36v2, EQ-5D, Work and Productivity Activity Impairment-Crohn's Disease (WPAI-CD) and disability.

It is estimated that approximately 800 subjects will be enrolled in total. All subjects will enter the study at baseline (Week 0) and commence oral treatment with GSK1605786A 500 mg twice daily.

The study will be conducted for 108 weeks. Once the results of the induction study CCX114151 are known, the risk-to-benefit ratio will be re-assessed and the study duration may be amended.

Study assessments for Crohn's disease will be performed every 12 weeks through Week 108. At week 12, the investigator will make a determination of whether the subject is receiving clinical benefit, and subjects who are not receiving clinical benefit must be withdrawn. More frequent blood draws are required for liver function testing only; every 2 weeks for the first 12 weeks, then every 4 weeks up to Week 52, and every 12 weeks after Week 60 for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in a GSK-sponsored study with GSK1605786A
* Written informed consent prior to any study-specific procedures
* Female subjects: To be eligible, females of child-bearing potential must be sexually inactive or commit to consistent and correct use of a contraceptive method of birth control with less than 1% failure rate

Exclusion Criteria:

* If female, is pregnant, has a positive pregnancy test or is breast-feeding, or is planning to become pregnant
* Subjects with known or suspected coeliac disease or a positive screening test for anti-tissue transglutaminase antibodies should have been excluded from enrolment into any induction study. Subjects in whom a diagnosis of coeliac disease is subsequently suspected should be tested for anti-tissue transglutaminase antibodies and excluded or withdrawn from the study upon positive test result
* Fixed symptomatic stenoses or strictures of small bowel or colon
* Enterocutaneous, abdominal or pelvic fistulae likely to require surgery during the study period
* Current sepsis or infections requiring intravenous antibiotic therapy greater than 2 weeks
* Evidence of hepatic dysfunction or viral hepatitis
* Subjects who have demonstrated safety or tolerability issues during participation in a previous study with GSK1605786A which, in the opinion of the investigator, was possibly related to study treatment and poses an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2011-04-01; Primary Completion 2013-09-01 (Actual); Study Completion 2013-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (206):
- United States (52):
  - GSK Investigational Site, Little Rock, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Hammond, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Lee's Summit, Missouri
  - GSK Investigational Site, Mexico, Missouri
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, East Setauket, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (8):
  - GSK Investigational Site, Bankstown, New South Wales
  - GSK Investigational Site, Hersten, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Kurralta Park, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Austria (5):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Oberpullendorf
  - GSK Investigational Site, St.Veit/Glan
  - GSK Investigational Site, Vienna
- Belgium (6):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (12):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Abbotsford, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Viña del Mar, Chile
- Czechia (4):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Vitkovice
  - GSK Investigational Site, Prague
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (8):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin, New Territories
- Hungary (6):
  - GSK Investigational Site, Békéscsaba
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Szekszárd
  - GSK Investigational Site, Vác
- Israel (10):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Ẕerifin
- Italy (4):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Roma
- Japan (10):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- New Zealand (4):
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Otahuhu, Auckland
  - GSK Investigational Site, Tauranga
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Wroclaw
- Portugal (3):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Viseu
- Russia (8):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tomsk
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Trnava
- South Africa (4):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Parktown
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wŏnju
- Spain (7):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Fuenlabrada (Madrid)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Santander
- Sweden (2):
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Switzerland (2):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Zurich
- GSK Investigational Site, Taichung, Taiwan
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- Ukraine (8):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
- United Kingdom (8):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible to enter the study if they completed the placebo-controlled induction study CCX114151; completed the maintenance study CCX114157 at Week 52; or withdrew from the maintenance study CCX114157. A total of such 800 participants were planned to be enrolled.
Pre-assignment Details: All participants entered the study at a Baseline visit, Week 0, and received GSK1605786A 500 milligrams (mg), twice daily (BID) for 216 weeks.
Groups:
- GSK1605786A: Eligible participants received oral GSK1605786A 500 mg BID for 216 weeks and were followed-up till 220 weeks. The participants who prematurely discontinued the study were followed by for last 4 weeks after receiving the last dose of the study drug.
Period: Overall Study
Arm/Group | GSK1605786A
Started | 398
Completed | 0
Not Completed | 398
Not completed — Adverse Event | 53
Not completed — Lack of Efficacy | 121
Not completed — Protocol Violation | 3
Not completed — Protocol based stopping criteria | 6
Not completed — Study closed or terminated | 174
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 13
Not completed — Withdrawal by Subject | 24

BASELINE CHARACTERISTICS:
Population: The safety population included all the participants who received at least one dose of the study drug.
Groups:
- GSK1605786A 500 mg BID: Eligible participants received oral GSK1605786A 500 mg BID for 216 weeks and were followed-up till 220 weeks. The participants who prematurely discontinued the study were followed by for last 4 weeks after receiving the last dose of the study drug.
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 351
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AE) and Any Serious Adverse Events (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; was a congenital anomaly/birth defect. The Safety population consisted of all participants who enrolled in the study except those who did not take >=1 dose of investigational product.
Time Frame: Up to Week 112
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Participants
  Any AE | 303
  Any SAE | 41

2. Secondary Outcome: Change From Baseline (Week 0) in Systolic and Diastolic Blood Pressure (SBP and DBP) Over Period
Description: The SBP and DBP values were obtained as part of vital sign monitoring and measured after the participant was at rest in the supine position for at least 5 minutes. Baseline value was recorded at Week 0. Change from Baseline measurements in SBP and DBP were assessed at Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 4 weeks post-treatment. The Baseline value is defined as the value at Week 0. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
millimeters of mercury (mmHg)
  SBP, Week 4: number analyzed (Participants) | 390
  SBP, Week 4 | -0.4 (11.39)
  SBP, Week 8: number analyzed (Participants) | 337
  SBP, Week 8 | -0.4 (11.46)
  SBP, Week 12: number analyzed (Participants) | 291
  SBP, Week 12 | -0.9 (13.12)
  SBP, Week 24: number analyzed (Participants) | 197
  SBP, Week 24 | 1.0 (12.69)
  SBP, Week 36: number analyzed (Participants) | 132
  SBP, Week 36 | 1.3 (12.64)
  SBP, Week 48: number analyzed (Participants) | 91
  SBP, Week 48 | -0.5 (13.22)
  SBP, Week 60: number analyzed (Participants) | 56
  SBP, Week 60 | 1.5 (13.00)
  SBP, Week 72: number analyzed (Participants) | 36
  SBP, Week 72 | -0.1 (13.15)
  SBP, Week 84: number analyzed (Participants) | 19
  SBP, Week 84 | 5.4 (18.65)
  SBP, Week 96: number analyzed (Participants) | 13
  SBP, Week 96 | -5.4 (10.72)
  SBP, Week 108: number analyzed (Participants) | 6
  SBP, Week 108 | 2.2 (13.44)
  SBP, 4 week post treatment: number analyzed (Participants) | 298
  SBP, 4 week post treatment | 0.5 (13.56)
  DBP, Week 4: number analyzed (Participants) | 390
  DBP, Week 4 | 0.1 (8.58)
  DBP, Week 8: number analyzed (Participants) | 337
  DBP, Week 8 | 0.1 (8.18)
  DBP, Week 12: number analyzed (Participants) | 291
  DBP, Week 12 | 0.2 (9.21)
  DBP, Week 24: number analyzed (Participants) | 197
  DBP, Week 24 | 0.1 (10.17)
  DBP, Week 36: number analyzed (Participants) | 132
  DBP, Week 36 | 1.0 (9.80)
  DBP, Week 48: number analyzed (Participants) | 91
  DBP, Week 48 | 0.0 (9.02)
  DBP, Week 60: number analyzed (Participants) | 56
  DBP, Week 60 | 1.2 (10.59)
  DBP, Week 72: number analyzed (Participants) | 36
  DBP, Week 72 | 0.0 (10.03)
  DBP, Week 84: number analyzed (Participants) | 19
  DBP, Week 84 | 4.4 (11.00)
  DBP, Week 96: number analyzed (Participants) | 13
  DBP, Week 96 | -1.8 (9.33)
  DBP, Week 108, n=6: number analyzed (Participants) | 6
  DBP, Week 108, n=6 | 1.3 (9.52)
  DBP, 4 week post treatment: number analyzed (Participants) | 298
  DBP, 4 week post treatment | 0.1 (9.91)

3. Secondary Outcome: Change From Baseline (Week 0) in Heart Rate (HR) Over Period
Description: The HR values were obtained as part of vital sign monitoring and measured after the participant was at rest in the supine position for at least 5 minutes. Change from Baseline in HR was assessed at Week 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 4 weeks post-treatment. The Baseline value is defined as the value at Week 0. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline (week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
beats per minute
  HR, Week 4: number analyzed (Participants) | 390
  HR, Week 4 | 1.3 (10.92)
  HR, Week 8: number analyzed (Participants) | 337
  HR, Week 8 | 0.1 (11.41)
  HR, Week 12: number analyzed (Participants) | 291
  HR, Week 12 | 0.8 (11.93)
  HR, Week 24: number analyzed (Participants) | 197
  HR, Week 24 | -0.5 (12.56)
  HR, Week 36: number analyzed (Participants) | 132
  HR, Week 36 | 2.1 (12.35)
  HR, Week 48: number analyzed (Participants) | 91
  HR, Week 48 | -1.2 (13.16)
  HR, Week 60: number analyzed (Participants) | 56
  HR, Week 60 | 0.4 (12.85)
  HR, Week 72: number analyzed (Participants) | 36
  HR, Week 72 | -1.2 (12.39)
  HR, Week 84: number analyzed (Participants) | 19
  HR, Week 84 | -0.7 (15.44)
  HR, Week 96: number analyzed (Participants) | 13
  HR, Week 96 | -4.9 (17.01)
  HR, Week 108: number analyzed (Participants) | 6
  HR, Week 108 | -7.7 (12.83)
  HR, 4 week post treatment: number analyzed (Participants) | 298
  HR, 4 week post treatment | -0.8 (12.89)

4. Secondary Outcome: Number of Participants With Shifts From Baseline (Week 0) for the Indicated Hematology Parameters
Description: Hematology parameters measured included platelets, neutrophils (NL), lymphocytes, monocytes, eosinophils, basophils, hematocrit, band cells, red blood cell (RBC) count, hemoglobin, white blood cell (WBC) count, and segmented (seg) NL. The Baseline value is defined as the value obtained at Week 0. The number of participants with the indicated hematology parameters data reference range shifts from Baseline (defined as shift to low, shift to normal or no change, shift to high) until 4 weeks post treatment are presented.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only the participants available at the time of analysis were included.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Participants
  Platelets, shift to low: number analyzed (Participants) | 393
  Platelets, shift to low | 2
  Platelets, shift to normal or no change: number analyzed (Participants) | 394
  Platelets, shift to normal or no change | 325
  Platelets, shift to high: number analyzed (Participants) | 295
  Platelets, shift to high | 67
  NL, shift to low: number analyzed (Participants) | 393
  NL, shift to low | 5
  NL, shift to normal or no change: number analyzed (Participants) | 395
  NL, shift to normal or no change | 284
  NL, shift to high: number analyzed (Participants) | 214
  NL, shift to high | 106
  Lymphocytes, shift to low: number analyzed (Participants) | 239
  Lymphocytes, shift to low | 99
  Lymphocytes, shift to normal or no change: number analyzed (Participants) | 395
  Lymphocytes, shift to normal or no change | 292
  Lymphocytes, shift to high: number analyzed (Participants) | 392
  Lymphocytes, shift to high | 4
  Monocytes, shift to low: number analyzed (Participants) | 395
  Monocytes, shift to low | 0
  Monocytes, shift to normal or no change: number analyzed (Participants) | 395
  Monocytes, shift to normal or no change | 372
  Monocytes, shift to high: number analyzed (Participants) | 383
  Monocytes, shift to high | 23
  Eosinophils, shift to normal or no change: number analyzed (Participants) | 395
  Eosinophils, shift to normal or no change | 366
  Eosinophils, shift to high: number analyzed (Participants) | 382
  Eosinophils, shift to high | 29
  Basophils, shift to normal or no change: number analyzed (Participants) | 395
  Basophils, shift to normal or no change | 395
  Basophils, shift to high: number analyzed (Participants) | 394
  Basophils, shift to high | 0
  Hematocrit, shift to low: number analyzed (Participants) | 249
  Hematocrit, shift to low | 75
  Hematocrit, shift to normal or no change: number analyzed (Participants) | 395
  Hematocrit, shift to normal or no change | 312
  Hematocrit, shift to high: number analyzed (Participants) | 392
  Hematocrit, shift to high | 8
  Band cells, shift to normal or no change: number analyzed (Participants) | 6
  Band cells, shift to normal or no change | 5
  Band cells, shift to high: number analyzed (Participants) | 2
  Band cells, shift to high | 1
  RBC Count, shift to low: number analyzed (Participants) | 293
  RBC Count, shift to low | 62
  RBC Count, shift to normal or no change: number analyzed (Participants) | 395
  RBC Count, shift to normal or no change | 322
  RBC Count, shift to high: number analyzed (Participants) | 393
  RBC Count, shift to high | 11
  Hemoglobin, shift to low: number analyzed (Participants) | 191
  Hemoglobin, shift to low | 74
  Hemoglobin, shift to normal or no change: number analyzed (Participants) | 395
  Hemoglobin, shift to normal or no change | 320
  Hemoglobin, shift to high: number analyzed (Participants) | 395
  Hemoglobin, shift to high | 1
  WBC Count, shift to low: number analyzed (Participants) | 388
  WBC Count, shift to low | 23
  WBC Count, shift to normal or no change: number analyzed (Participants) | 395
  WBC Count, shift to normal or no change | 289
  WBC Count, shift to high: number analyzed (Participants) | 313
  WBC Count, shift to high | 83
  Segmented (Seg) NL, shift to low: number analyzed (Participants) | 393
  Segmented (Seg) NL, shift to low | 5
  Seg NL, shift to normal or no change: number analyzed (Participants) | 395
  Seg NL, shift to normal or no change | 283
  Seg NL, shift to high: number analyzed (Participants) | 215
  Seg NL, shift to high | 107

5. Secondary Outcome: Number of Participants With Shifts From Baseline (Week 0) for the Indicated Clinical Chemistry Parameters
Description: Clinical chemistry parameters included platelets, total protein, phosphorous, albumin, sodium, potassium, chloride, calcium, glucose, gamma-glutamyl transferase, total bilirubin (TB), direct bilirubin (DB), alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN)/urea, creatinine, uric acid, bicarbonate, lactate dehydrogenase, cholesterol, alkaline phosphatase (ALP), gamma glutamyl transferases (GGT), and creatine kinase. The Baseline value is defined as the value obtained at Week 0. The number of participants with the indicated clinical chemistry parameters' data reference range shifts from Baseline (defined as shift to low, shift to normal or no change, or shift to high) until 4 weeks post-treatment are presented.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Participants
  Total Protein, shift to low: number analyzed (Participants) | 370
  Total Protein, shift to low | 27
  Total Protein, shift to normal or no change: number analyzed (Participants) | 395
  Total Protein, shift to normal or no change | 367
  Total Protein, shift to high: number analyzed (Participants) | 395
  Total Protein, shift to high | 1
  Phosphorous, shift to low: number analyzed (Participants) | 369
  Phosphorous, shift to low | 85
  Phosphorous, shift to normal or no change: number analyzed (Participants) | 395
  Phosphorous, shift to normal or no change | 283
  Phosphorous, shift to high: number analyzed (Participants) | 385
  Phosphorous, shift to high | 30
  Albumin, shift to low: number analyzed (Participants) | 372
  Albumin, shift to low | 19
  Albumin, shift to normal or no change: number analyzed (Participants) | 395
  Albumin, shift to normal or no change | 373
  Albumin, shift to high: number analyzed (Participants) | 395
  Albumin, shift to high | 3
  Sodium, shift to low: number analyzed (Participants) | 392
  Sodium, shift to low | 18
  Sodium, shift to normal or no change: number analyzed (Participants) | 395
  Sodium, shift to normal or no change | 376
  Sodium, shift to high: number analyzed (Participants) | 395
  Sodium, shift to high | 1
  Potassium, shift to low: number analyzed (Participants) | 379
  Potassium, shift to low | 25
  Potassium, shift to normal or no change: number analyzed (Participants) | 395
  Potassium, shift to normal or no change | 360
  Potassium, shift to high: number analyzed (Participants) | 393
  Potassium, shift to high | 10
  Chloride, shift to low: number analyzed (Participants) | 395
  Chloride, shift to low | 3
  Chloride, shift to normal or no change: number analyzed (Participants) | 395
  Chloride, shift to normal or no change | 361
  Chloride, shift to high: number analyzed (Participants) | 381
  Chloride, shift to high | 31
  Calcium, shift to low: number analyzed (Participants) | 363
  Calcium, shift to low | 43
  Calcium, shift to normal or no change: number analyzed (Participants) | 395
  Calcium, shift to normal or no change | 340
  Calcium, shift to high: number analyzed (Participants) | 394
  Calcium, shift to high | 12
  Glucose, shift to low: number analyzed (Participants) | 370
  Glucose, shift to low | 54
  Glucose, shift to normal or no change: number analyzed (Participants) | 395
  Glucose, shift to normal or no change | 279
  Glucose, shift to high: number analyzed (Participants) | 361
  Glucose, shift to high | 66
  GGT, shift to normal or no change: number analyzed (Participants) | 397
  GGT, shift to normal or no change | 330
  GGT, shift to high: number analyzed (Participants) | 355
  GGT, shift to high | 67
  TB, shift to normal or no change: number analyzed (Participants) | 397
  TB, shift to normal or no change | 391
  TB, shift to high: number analyzed (Participants) | 393
  TB, shift to high | 6
  DB, shift to normal or no change: number analyzed (Participants) | 397
  DB, shift to normal or no change | 397
  DB, shift to high: number analyzed (Participants) | 397
  DB, shift to high | 0
  ALP, shift to low: number analyzed (Participants) | 395
  ALP, shift to low | 0
  ALP, shift to normal or no change, n=397: number analyzed (Participants) | 397
  ALP, shift to normal or no change, n=397 | 357
  ALP, shift to high, n=370: number analyzed (Participants) | 370
  ALP, shift to high, n=370 | 14
  ALT, shift to low, n=0: number analyzed (Participants) | 0
  ALT, shift to normal or no change: number analyzed (Participants) | 397
  ALT, shift to normal or no change | 349
  ALT, shift to high: number analyzed (Participants) | 390
  ALT, shift to high | 48
  AST, shift to low: number analyzed (Participants) | 0
  AST, shift to normal or no change: number analyzed (Participants) | 397
  AST, shift to normal or no change | 362
  AST, shift to high: number analyzed (Participants) | 390
  AST, shift to high | 35
  BUN/Urea, shift to low: number analyzed (Participants) | 367
  BUN/Urea, shift to low | 44
  BUN/Urea, shift to normal or no change: number analyzed (Participants) | 395
  BUN/Urea, shift to normal or no change | 345
  BUN/Urea, shift to high: number analyzed (Participants) | 393
  BUN/Urea, shift to high | 6
  Creatinine, shift to low: number analyzed (Participants) | 326
  Creatinine, shift to low | 50
  Creatinine, shift to normal or no change: number analyzed (Participants) | 395
  Creatinine, shift to normal or no change | 335
  Creatinine, shift to high: number analyzed (Participants) | 392
  Creatinine, shift to high | 10
  Uric Acid, shift to low: number analyzed (Participants) | 382
  Uric Acid, shift to low | 21
  Uric Acid, shift to normal or no change: number analyzed (Participants) | 395
  Uric Acid, shift to normal or no change | 350
  Uric Acid, shift to high: number analyzed (Participants) | 390
  Uric Acid, shift to high | 24
  Bicarbonate, shift to low: number analyzed (Participants) | 355
  Bicarbonate, shift to low | 92
  Bicarbonate, shift to normal or no change: number analyzed (Participants) | 395
  Bicarbonate, shift to normal or no change | 303
  Bicarbonate, shift to high: number analyzed (Participants) | 394
  Bicarbonate, shift to high | 0
  LDH, shift to normal or no change: number analyzed (Participants) | 395
  LDH, shift to normal or no change | 386
  LDH, shift to high: number analyzed (Participants) | 392
  LDH, shift to high | 9
  Cholesterol, shift to normal or no change: number analyzed (Participants) | 395
  Cholesterol, shift to normal or no change | 330
  Cholesterol, shift to high: number analyzed (Participants) | 335
  Cholesterol, shift to high | 65
  CK, shift to normal or no change: number analyzed (Participants) | 395
  CK, shift to normal or no change | 357
  CK, shift to high: number analyzed (Participants) | 386
  CK, shift to high | 38

6. Secondary Outcome: Change From Baseline (Week 0) in ALT, AST, ALP, and GGT as a Function of Liver Function Test (LFT)
Description: Changes in Baseline in ALP, ALT, AST, and GGT were assessed to monitor liver function. Blood samples were taken at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72, 84, 96, 108, and 4 Weeks post-treatment. The last value on or prior to the treatment start date was considered the Baseline value. Change from Baseline was calculated as the post-Baseline value at the time point indicated minus the value at Baseline.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Unit per Liter (IU/L)
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
International Unit per Liter (IU/L)
  ALT, Week 2: number analyzed (Participants) | 374
  ALT, Week 2 | 15.2 (11.33)
  ALT, Week 4: number analyzed (Participants) | 365
  ALT, Week 4 | 19.3 (43.93)
  ALT, Week 6: number analyzed (Participants) | 348
  ALT, Week 6 | 17.0 (18.98)
  ALT, Week 8: number analyzed (Participants) | 322
  ALT, Week 8 | 17.0 (23.94)
  ALT, Week 10: number analyzed (Participants) | 297
  ALT, Week 10 | 16.1 (16.17)
  ALT, Week 12: number analyzed (Participants) | 281
  ALT, Week 12 | 16.7 (17.07)
  ALT, Week 16: number analyzed (Participants) | 229
  ALT, Week 16 | 16.2 (13.77)
  ALT, Week 20: number analyzed (Participants) | 203
  ALT, Week 20 | 17.9 (32.94)
  ALT, Week 24: number analyzed (Participants) | 182
  ALT, Week 24 | 15.2 (10.77)
  ALT, Week 28: number analyzed (Participants) | 158
  ALT, Week 28 | 17.1 (20.11)
  ALT, Week 32: number analyzed (Participants) | 141
  ALT, Week 32 | 15.7 (12.25)
  ALT, Week 36: number analyzed (Participants) | 121
  ALT, Week 36 | 15.8 (10.74)
  ALT, Week 40: number analyzed (Participants) | 102
  ALT, Week 40 | 16.6 (11.49)
  ALT, Week 44: number analyzed (Participants) | 95
  ALT, Week 44 | 17.4 (12.77)
  ALT, Week 48: number analyzed (Participants) | 89
  ALT, Week 48 | 15.0 (7.61)
  ALT, Week 52: number analyzed (Participants) | 77
  ALT, Week 52 | 14.7 (7.74)
  ALT, Week 60: number analyzed (Participants) | 55
  ALT, Week 60 | 16.0 (10.20)
  ALT, Week 72: number analyzed (Participants) | 36
  ALT, Week 72 | 15.1 (6.55)
  ALT, Week 84: number analyzed (Participants) | 18
  ALT, Week 84 | 15.4 (7.11)
  ALT, Week 96: number analyzed (Participants) | 13
  ALT, Week 96 | 16.8 (6.03)
  ALT, Week 108: number analyzed (Participants) | 6
  ALT, Week 108 | 15.7 (7.69)
  ALT, 4 week post treatment: number analyzed (Participants) | 299
  ALT, 4 week post treatment | 18.9 (22.52)
  AST, Week 2: number analyzed (Participants) | 373
  AST, Week 2 | 16.9 (6.87)
  AST, Week 4: number analyzed (Participants) | 365
  AST, Week 4 | 18.6 (19.31)
  AST, Week 6: number analyzed (Participants) | 348
  AST, Week 6 | 17.6 (9.56)
  AST, Week 8: number analyzed (Participants) | 322
  AST, Week 8 | 17.7 (14.11)
  AST, Week 10: number analyzed (Participants) | 296
  AST, Week 10 | 17.4 (9.51)
  AST, Week 12: number analyzed (Participants) | 280
  AST, Week 12 | 19.2 (25.75)
  AST, Week 16: number analyzed (Participants) | 228
  AST, Week 16 | 17.8 (8.76)
  AST, Week 20: number analyzed (Participants) | 202
  AST, Week 20 | 19.4 (21.90)
  AST, Week 24: number analyzed (Participants) | 182
  AST, Week 24 | 17.8 (7.92)
  AST, Week 28: number analyzed (Participants) | 158
  AST, Week 28 | 18.6 (12.59)
  AST, Week 32: number analyzed (Participants) | 141
  AST, Week 32 | 18.1 (8.55)
  AST, Week 36: number analyzed (Participants) | 120
  AST, Week 36 | 18.4 (8.01)
  AST, Week 40: number analyzed (Participants) | 102
  AST, Week 40 | 18.4 (7.68)
  AST, Week 44: number analyzed (Participants) | 95
  AST, Week 44 | 18.7 (8.66)
  AST, Week 48: number analyzed (Participants) | 89
  AST, Week 48 | 17.6 (6.11)
  AST, Week 52: number analyzed (Participants) | 77
  AST, Week 52 | 17.1 (5.71)
  AST, Week 60: number analyzed (Participants) | 55
  AST, Week 60 | 18.4 (6.07)
  AST, Week 72: number analyzed (Participants) | 36
  AST, Week 72 | 17.2 (3.80)
  AST, Week 84: number analyzed (Participants) | 18
  AST, Week 84 | 18.2 (4.96)
  AST, Week 96: number analyzed (Participants) | 13
  AST, Week 96 | 19.7 (5.92)
  AST, Week 108: number analyzed (Participants) | 6
  AST, Week 108 | 18.2 (4.22)
  AST, 4 week post treatment: number analyzed (Participants) | 298
  AST, 4 week post treatment | 19.6 (13.82)
  ALP, Week 2: number analyzed (Participants) | 374
  ALP, Week 2 | 81.1 (26.52)
  ALP, Week 4: number analyzed (Participants) | 365
  ALP, Week 4 | 82.3 (27.61)
  ALP, Week 6: number analyzed (Participants) | 348
  ALP, Week 6 | 82.0 (27.46)
  ALP, Week 8: number analyzed (Participants) | 322
  ALP, Week 8 | 81.3 (25.60)
  ALP, Week 10: number analyzed (Participants) | 297
  ALP, Week 10 | 81.3 (25.60)
  ALP, Week 12: number analyzed (Participants) | 281
  ALP, Week 12 | 81.1 (26.31)
  ALP, Week 16: number analyzed (Participants) | 229
  ALP, Week 16 | 80.8 (26.50)
  ALP, Week 20: number analyzed (Participants) | 203
  ALP, Week 20 | 80.8 (22.68)
  ALP, Week 24: number analyzed (Participants) | 182
  ALP, Week 24 | 83.4 (23.51)
  ALP, Week 28: number analyzed (Participants) | 158
  ALP, Week 28 | 83.3 (25.45)
  ALP, Week 32: number analyzed (Participants) | 141
  ALP, Week 32 | 84.5 (25.03)
  ALP, Week 36: number analyzed (Participants) | 121
  ALP, Week 36 | 83.8 (24.89)
  ALP, Week 40: number analyzed (Participants) | 102
  ALP, Week 40 | 82.8 (22.31)
  ALP, Week 44: number analyzed (Participants) | 95
  ALP, Week 44 | 81.5 (20.35)
  ALP, Week 48: number analyzed (Participants) | 89
  ALP, Week 48 | 81.5 (25.02)
  ALP, Week 52: number analyzed (Participants) | 77
  ALP, Week 52 | 79.0 (18.80)
  ALP, Week 60: number analyzed (Participants) | 55
  ALP, Week 60 | 78.9 (20.55)
  ALP, Week 72: number analyzed (Participants) | 36
  ALP, Week 72 | 78.1 (19.76)
  ALP, Week 84: number analyzed (Participants) | 18
  ALP, Week 84 | 78.4 (21.76)
  ALP, Week 96: number analyzed (Participants) | 13
  ALP, Week 96 | 78.2 (20.67)
  ALP, Week 108: number analyzed (Participants) | 6
  ALP, Week 108 | 81.5 (19.64)
  ALP, 4 week post treatment: number analyzed (Participants) | 299
  ALP, 4 week post treatment | 82.7 (31.50)
  GGT, Week 2: number analyzed (Participants) | 374
  GGT, Week 2 | 31.2 (23.61)
  GGT, Week 4: number analyzed (Participants) | 365
  GGT, Week 4 | 34.0 (32.84)
  GGT, Week 6: number analyzed (Participants) | 347
  GGT, Week 6 | 32.9 (28.44)
  GGT, Week 8: number analyzed (Participants) | 322
  GGT, Week 8 | 32.6 (24.78)
  GGT, Week 10: number analyzed (Participants) | 297
  GGT, Week 10 | 31.7 (26.63)
  GGT, Week 12: number analyzed (Participants) | 281
  GGT, Week 12 | 33.0 (29.49)
  GGT, Week 16: number analyzed (Participants) | 229
  GGT, Week 16 | 32.3 (28.17)
  GGT, Week 20: number analyzed (Participants) | 203
  GGT, Week 20 | 32.3 (26.99)
  GGT, Week 24: number analyzed (Participants) | 182
  GGT, Week 24 | 33.5 (30.74)
  GGT, Week 28: number analyzed (Participants) | 158
  GGT, Week 28 | 35.2 (34.85)
  GGT, Week 32: number analyzed (Participants) | 141
  GGT, Week 32 | 35.1 (31.75)
  GGT, Week 36: number analyzed (Participants) | 121
  GGT, Week 36 | 34.0 (29.18)
  GGT, Week 40: number analyzed (Participants) | 102
  GGT, Week 40 | 34.2 (29.22)
  GGT, Week 44: number analyzed (Participants) | 95
  GGT, Week 44 | 30.9 (19.33)
  GGT, Week 48: number analyzed (Participants) | 89
  GGT, Week 48 | 31.6 (29.92)
  GGT, Week 52: number analyzed (Participants) | 77
  GGT, Week 52 | 29.3 (18.45)
  GGT, Week 60: number analyzed (Participants) | 55
  GGT, Week 60 | 32.6 (23.50)
  GGT, Week 72: number analyzed (Participants) | 36
  GGT, Week 72 | 32.2 (25.30)
  GGT, Week 84: number analyzed (Participants) | 18
  GGT, Week 84 | 33.7 (28.66)
  GGT, Week 96: number analyzed (Participants) | 13
  GGT, Week 96 | 34.1 (29.97)
  GGT, Week 108: number analyzed (Participants) | 6
  GGT, Week 108 | 24.5 (11.62)
  GGT, 4 week post treatment: number analyzed (Participants) | 297
  GGT, 4 week post treatment | 31.7 (30.19)

7. Secondary Outcome: Change From Baseline (Week 0) in Total Bilirubin
Description: Changes from Baseline (Week 0) in total bilirubin (TB) was assessed to monitor liver function. Blood samples were taken at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72, 84, 96, 108, and 4 Weeks post-treatment. The last value on or prior to the treatment start date was considered the Baseline value. Change from Baseline was calculated as the post-Baseline value at the time point indicated minus the value at Baseline.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
micromole/Liter
  TB, Week 2: number analyzed (Participants) | 374
  TB, Week 2 | 6.9 (2.85)
  TB, Week 4: number analyzed (Participants) | 365
  TB, Week 4 | 7.1 (3.24)
  TB, Week 6: number analyzed (Participants) | 348
  TB, Week 6 | 6.8 (2.76)
  TB, Week 8: number analyzed (Participants) | 322
  TB, Week 8 | 6.8 (2.61)
  TB, Week 10: number analyzed (Participants) | 297
  TB, Week 10 | 7.1 (2.91)
  TB, Week 12: number analyzed (Participants) | 281
  TB, Week 12 | 6.7 (2.54)
  TB, Week 16: number analyzed (Participants) | 229
  TB, Week 16 | 7.0 (2.78)
  TB, Week 20: number analyzed (Participants) | 203
  TB, Week 20 | 6.9 (2.99)
  TB, Week 24: number analyzed (Participants) | 182
  TB, Week 24 | 7.2 (2.80)
  TB, Week 28: number analyzed (Participants) | 158
  TB, Week 28 | 7.0 (2.70)
  TB, Week 32: number analyzed (Participants) | 141
  TB, Week 32 | 6.9 (2.58)
  TB, Week 36: number analyzed (Participants) | 121
  TB, Week 36 | 7.1 (2.42)
  TB, Week 40: number analyzed (Participants) | 102
  TB, Week 40 | 7.4 (3.01)
  TB, Week 44: number analyzed (Participants) | 95
  TB, Week 44 | 7.4 (2.56)
  TB, Week 48: number analyzed (Participants) | 89
  TB, Week 48 | 7.0 (2.35)
  TB, Week 52: number analyzed (Participants) | 77
  TB, Week 52 | 7.0 (2.57)
  TB, Week 60: number analyzed (Participants) | 55
  TB, Week 60 | 7.3 (2.05)
  TB, Week 72: number analyzed (Participants) | 36
  TB, Week 72 | 7.1 (2.38)
  TB, Week 84: number analyzed (Participants) | 18
  TB, Week 84 | 7.2 (2.44)
  TB, Week 96: number analyzed (Participants) | 13
  TB, Week 96 | 8.1 (2.29)
  TB, Week 108: number analyzed (Participants) | 6
  TB, Week 108 | 7.0 (1.79)
  TB, 4 week post treatment: number analyzed (Participants) | 299
  TB, 4 week post treatment | 8.4 (4.11)

8. Secondary Outcome: Change From Baseline (Week 0) in Albumin
Description: Change from Baseline in albumin was assessed to monitor liver function. Blood samples were taken at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, 72, 84, 96, 108, and 4 Weeks post treatment. The last value on or prior to the treatment start date (Week 0) was considered the Baseline value. Change from Baseline was calculated as the post-Baseline value at the time point indicated minus the value at Baseline.
Time Frame: Baseline (Week 0) and up to Week 112
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams/Liter (G/L)
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Grams/Liter (G/L)
  Albumin, Week 2: number analyzed (Participants) | 20
  Albumin, Week 2 | 39.4 (5.68)
  Albumin, Week 4: number analyzed (Participants) | 356
  Albumin, Week 4 | 39.8 (4.76)
  Albumin, Week 6: number analyzed (Participants) | 31
  Albumin, Week 6 | 40.4 (4.88)
  Albumin, Week 8: number analyzed (Participants) | 317
  Albumin, Week 8 | 40.0 (4.80)
  Albumin, Week 10: number analyzed (Participants) | 19
  Albumin, Week 10 | 40.5 (4.94)
  Albumin, Week 12: number analyzed (Participants) | 277
  Albumin, Week 12 | 40.3 (4.56)
  Albumin, Week 16: number analyzed (Participants) | 22
  Albumin, Week 16 | 37.9 (5.40)
  Albumin, Week 20: number analyzed (Participants) | 19
  Albumin, Week 20 | 42.2 (3.30)
  Albumin, Week 24: number analyzed (Participants) | 181
  Albumin, Week 24 | 41.0 (4.28)
  Albumin, Week 28: number analyzed (Participants) | 8
  Albumin, Week 28 | 40.1 (5.54)
  Albumin, Week 32: number analyzed (Participants) | 8
  Albumin, Week 32 | 35.8 (8.01)
  Albumin, Week 36: number analyzed (Participants) | 121
  Albumin, Week 36 | 41.4 (4.81)
  Albumin, Week 40: number analyzed (Participants) | 6
  Albumin, Week 40 | 41.5 (3.02)
  Albumin, Week 44: number analyzed (Participants) | 1
  Albumin, Week 44 | 41.0 (NA) — SD could not be calculated since only 1 participant was analyzed.
  Albumin, Week 48: number analyzed (Participants) | 88
  Albumin, Week 48 | 41.0 (5.22)
  Albumin, Week 52: number analyzed (Participants) | 6
  Albumin, Week 52 | 41.3 (6.22)
  Albumin, Week 60: number analyzed (Participants) | 55
  Albumin, Week 60 | 41.4 (4.38)
  Albumin, Week 72: number analyzed (Participants) | 36
  Albumin, Week 72 | 42.0 (4.89)
  Albumin, Week 84: number analyzed (Participants) | 18
  Albumin, Week 84 | 41.9 (4.20)
  Albumin, Week 96: number analyzed (Participants) | 13
  Albumin, Week 96 | 43.2 (2.28)
  Albumin, Week 108: number analyzed (Participants) | 6
  Albumin, Week 108 | 44.7 (3.72)
  Albumin, 4 week post treatment: number analyzed (Participants) | 295
  Albumin, 4 week post treatment | 40.6 (4.46)

9. Secondary Outcome: Number of Participants With the Indicated Change From Baseline (Week 0) in Corrected QT Interval (QTc) Value
Description: QTc is the corrected QT interval as measured by the electrocardiogram (ECG). ECG parameters including the change from Baseline in the QTc interval values QTcF and QTcB were summarised. The QTcF is Fridericia's formula and defined as the QT interval/cubed root of the R-R interval. The QTcB is the Bazett's formula defined as the QT/squared root of the R-R interval. The number of participants with change from Baseline in the QTcF and QTcB intervals of >30, 30 to <60 and >=60 milliseconds were assessed at Week 24, 48, 72, 108, and Week 112. The last value on or prior to the treatment start date was considered the Baseline value (Week 0). Change from Baseline was calculated as the post-Baseline value minus the value at Baseline.
Time Frame: Baseline (week 0) and Weeks 24, 48, 72, 108, and 112 (4 weeks post treatment)
Population: Safety Population. Only participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Participants
  QTcB, Week 24,<30, n=70: number analyzed (Participants) | 70
  QTcB, Week 24,<30, n=70 | 66
  QTcB, Week 24, 30-<60, n=70: number analyzed (Participants) | 70
  QTcB, Week 24, 30-<60, n=70 | 3
  QTcB, Week 24, >=60, n=70: number analyzed (Participants) | 70
  QTcB, Week 24, >=60, n=70 | 1
  QTcB, Week 48,<30, n=35: number analyzed (Participants) | 35
  QTcB, Week 48,<30, n=35 | 34
  QTcB, Week 48, 30-<60, n=35: number analyzed (Participants) | 35
  QTcB, Week 48, 30-<60, n=35 | 0
  QTcB, Week 48, >=60, n=35: number analyzed (Participants) | 35
  QTcB, Week 48, >=60, n=35 | 1
  QTcB, Week 72,<30, n=17: number analyzed (Participants) | 17
  QTcB, Week 72,<30, n=17 | 15
  QTcB, Week 72, 30-<60, n=17: number analyzed (Participants) | 17
  QTcB, Week 72, 30-<60, n=17 | 1
  QTcB, Week 72, >=60, n=17: number analyzed (Participants) | 17
  QTcB, Week 72, >=60, n=17 | 1
  QTcB, Week 108,<30, n=3: number analyzed (Participants) | 3
  QTcB, Week 108,<30, n=3 | 3
  QTcB, Week 108, 30-<60, n=3: number analyzed (Participants) | 3
  QTcB, Week 108, 30-<60, n=3 | 0
  QTcB, Week 108, >=60, n=3: number analyzed (Participants) | 3
  QTcB, Week 108, >=60, n=3 | 0
  QTcB, 4 Weeks Post Treatment, <30, n=96: number analyzed (Participants) | 96
  QTcB, 4 Weeks Post Treatment, <30, n=96 | 89
  QTcB, 4 Weeks Post Treatment, 30-<60, n=96: number analyzed (Participants) | 96
  QTcB, 4 Weeks Post Treatment, 30-<60, n=96 | 6
  QTcB, 4 Weeks Post Treatment, >=60, n=96: number analyzed (Participants) | 96
  QTcB, 4 Weeks Post Treatment, >=60, n=96 | 1
  QTcF, Week 24,<30, n=23: number analyzed (Participants) | 23
  QTcF, Week 24,<30, n=23 | 22
  QTcF, Week 24, 30-<60, n=23: number analyzed (Participants) | 23
  QTcF, Week 24, 30-<60, n=23 | 1
  QTcF, Week 24, >=60, n=23: number analyzed (Participants) | 23
  QTcF, Week 24, >=60, n=23 | 0
  QTcF, Week 48,<30, n=13: number analyzed (Participants) | 13
  QTcF, Week 48,<30, n=13 | 13
  QTcF, Week 48, 30-<60, n=13: number analyzed (Participants) | 13
  QTcF, Week 48, 30-<60, n=13 | 0
  QTcB, Week 48, >=60, n=13: number analyzed (Participants) | 13
  QTcB, Week 48, >=60, n=13 | 0
  QTcF, Week 72,<30, n=7: number analyzed (Participants) | 7
  QTcF, Week 72,<30, n=7 | 7
  QTcF, Week 72, 30-<60, n=7: number analyzed (Participants) | 7
  QTcF, Week 72, 30-<60, n=7 | 0
  QTcF, Week 72, >=60, n=7: number analyzed (Participants) | 7
  QTcF, Week 72, >=60, n=7 | 0
  QTcF, Week 108,<30, n=2: number analyzed (Participants) | 2
  QTcF, Week 108,<30, n=2 | 1
  QTcF, Week 108, 30-<60, n=2: number analyzed (Participants) | 2
  QTcF, Week 108, 30-<60, n=2 | 1
  QTcF, Week 108, >=60, n=2: number analyzed (Participants) | 2
  QTcF, Week 108, >=60, n=2 | 0
  QTcF, 4 Weeks Post Treatment, <30, n=32: number analyzed (Participants) | 32
  QTcF, 4 Weeks Post Treatment, <30, n=32 | 32
  QTcF, 4 Weeks Post Treatment, 30-<60, n=32: number analyzed (Participants) | 32
  QTcF, 4 Weeks Post Treatment, 30-<60, n=32 | 0
  QTcF, 4 Weeks Post Treatment, >=60, n=32: number analyzed (Participants) | 32
  QTcF, 4 Weeks Post Treatment, >=60, n=32 | 0

10. Secondary Outcome: Change From Baseline (Week 0) in Crohn's Disease Activity Index (CDAI) Score Over 108 Weeks
Description: The CDAI score was determined by interactive voice response relationship (IVRS) based on the combination of participant,investigator entries, standardized weight determination, and Hematocrit values received from the central laboratory. The Baseline CDAI score was recorded pre-dose on Week 0. Change from Baseline is the value at indicated time point minus the Baseline value. Remissions are defined as participants with CDAI score of < 150 points. No imputation for missing data was performed. The assessment was based on questionnaire like number of liquid stool in past 7 days, abdominal pain, other symptoms, antidiarrheal use, abdominal mass, anemia, and body weight. The total score is summation of all individual sub-scores. CDAI scoring scale ranges from 0-500 and a score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Baseline (Week 0) and up to 108 weeks
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Scores on a scale
  Week 12: number analyzed (Participants) | 234
  Week 12 | -76.0 (92.79)
  Week 24: number analyzed (Participants) | 153
  Week 24 | -89.2 (102.87)
  Week 36: number analyzed (Participants) | 97
  Week 36 | -103.6 (113.63)
  Week 48: number analyzed (Participants) | 68
  Week 48 | -116.6 (109.42)
  Week 60: number analyzed (Participants) | 41
  Week 60 | -121.3 (111.29)
  Week 72: number analyzed (Participants) | 27
  Week 72 | -110.4 (104.18)
  Week 84: number analyzed (Participants) | 18
  Week 84 | -121.4 (115.70)
  Week 96: number analyzed (Participants) | 9
  Week 96 | -91.0 (80.00)
  Week 108: number analyzed (Participants) | 3
  Week 108 | -50.7 (19.86)

11. Secondary Outcome: Percentage of Participants in Clinical Remission (CDAI Score Less Than 150) for All Participants, for Participants in Remission at Baseline (Week 0), and for Participants Not in Remission at Baseline Over 108 Weeks
Description: The CDAI score was determined by interactive voice response relationship (IVRS) based on the combination of participant and investigator entries and standardized weight determination. Haematocrit values received from the central laboratory on the day of the visit were to be utilized for calculation of the CDAI scores. The Baseline (Week 0) CDAI score was defined as the last evaluation prior to or on the date the first dose of investigational product is taken. The CDAI score was measured over 108 weeks although it was planned to be measured till 112 weeks. Remissions are defined as subjects with CDAI score of < 150 points. Percentages are based on the number of subjects with observed data. No imputation for missing data was performed. Combined data for participants with remission at Baseline and without remission at Baseline has been presented.
Time Frame: Baseline (Week 0) and up to 108 weeks
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 398
Participants
  Week 0 | 8.5 [5.8 to 11.3]
  Week 12: number analyzed (Participants) | 234
  Week 12 | 35.0 [28.9 to 41.2]
  Week 24: number analyzed (Participants) | 153
  Week 24 | 41.2 [33.4 to 49.0]
  Week 36: number analyzed (Participants) | 97
  Week 36 | 52.6 [42.6 to 62.5]
  Week 48: number analyzed (Participants) | 68
  Week 48 | 54.4 [42.6 to 66.2]
  Week 60: number analyzed (Participants) | 41
  Week 60 | 53.7 [38.4 to 68.9]
  Week 72: number analyzed (Participants) | 27
  Week 72 | 51.9 [33.0 to 70.7]
  Week 84: number analyzed (Participants) | 18
  Week 84 | 55.6 [32.6 to 78.5]
  Week 96: number analyzed (Participants) | 9
  Week 96 | 66.7 [35.9 to 97.5]
  Week 108: number analyzed (Participants) | 3
  Week 108 | 33.3 [0.0 to 86.7]

12. Secondary Outcome: Percentage of Participants Achieving Response (CDAI Decrease of at Least 100 Points From Baseline ([Week 0] of Prior Induction Study) in the Sub-population of Non-responders at Study Entry Over 112 Weeks
Description: The CDAI score was determined by interactive voice response relationship (IVRS) based on the combination of participant and investigator entries and standardized weight determination. Haematocrit values received from the central laboratory on the day of the visit were to be utilized for calculation of the CDAI scores. The Baseline (Week 0) CDAI score was defined as the last evaluation prior to or on the date the first dose of investigational product was taken. Remissions are defined as subjects with CDAI score of < 150 points. Percentages are based on the number of subjects with observed data. No imputation for missing data was performed.
Time Frame: Baseline (Week 0) and up to 112 weeks
Population: ITT population was planned to be analyzed for this study.However, this outcome measure was not analyzed due to termination of study and no data was collected for this outcome measure.
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline (Week 0) in Inflammatory Bowel Disease Questionnaire (IBDQ), Short Form Health Survey (SF-36) Version 2, EuroQol 5 Dimensional (EQ-5D), Work and Productivity Activity Impairment-Crohn's Disease (WPAI-CD) and Disability Over 112 Weeks
Description: IBDQ, SF-36, EQ-5D, WPAI-CD, and disability scores were all health outcome related scores that were based on assessment of participants based on different questionnaire. Each scoring scale had different range and participants were planned to be rated separately based on each scale.
Time Frame: Baseline (Week 0) and up to 112 weeks
Population: ITT population was planned to be analyzed for this study. However, this outcome measure was not analyzed due to termination of study and no data was collected for this outcome measure.
Arm/Group | GSK1605786A 500 mg BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow-up visit (up to 112 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for members of the safety Population, comprised of all participants who enrolled in the study except those who did not take at least one dose of investigational product.
Arm/Group | GSK1605786A
All-Cause Mortality (participants affected / at risk) | 0/398
Serious Adverse Events (participants affected / at risk) | 41/398
Other Adverse Events (participants affected / at risk) | 295/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1605786A (N=398)
Crohn's disease (Gastrointestinal disorders) | 8
Anal fistula (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrointestinal stenosis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Anal abscess (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Shigella infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 3
Liver function test abnormal (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Drug ineffective (General disorders) | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Bartholinitis (Reproductive system and breast disorders) | 1
Intermittent claudication (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1605786A (N=398)
Headache (Nervous system disorders) | 42
Abdominal Pain (Gastrointestinal disorders) | 49
Crohn's Disease (Gastrointestinal disorders) | 49
Nausea (Gastrointestinal disorders) | 26
Diarrhea (Gastrointestinal disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Nasopharyngitis (Infections and infestations) | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.